CLINICAL TRIAL: NCT06751992
Title: Neurocognitive Function Changes With Once-Daily Extended-Release Tacrolimus (Envarsus XR) Conversion Compared to Twice-Daily Immediate Release Tacrolimus Maintenance Among Older Kidney Transplant Recipients
Brief Title: Neurocognitive Function Changes With Extended-Release Tacrolimus Among Older Kidney Transplant Recipients
Acronym: Neuro-KTR
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Veloxis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Leonardo V. Riella, MD, PhD, Medical Director of Kidney Transplantation, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2024P000460
Record Dates: First submitted 2024-12-13; First posted 2024-12-30 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Kidney Transplant Recipients; Old Age
Keywords: Neurocognitive function; Tacrolimus; Kidney transplant recipients; Tremor; Insomnia
MeSH Terms: conditions — Tremor; Sleep Initiation and Maintenance Disorders | interventions — Tacrolimus

STUDY DESIGN:
Intervention Model Description: A prospective, open-label, single-center, randomized controlled phase 4 trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Envarsus XR conversion (Experimental): Patients who are randomized to this group will receive extended-release tacrolimus (Envarsus XR) at 80 percent of their total daily dose of IR tacrolimus (Prograf) before the switch. Tacrolimus trough level will be obtained 3-4 weeks after the conversion to ensure appropriate dosage.
  Interventions: Drug: Conversion to extended-release tacrolimus
- Prograf maintenance (Active Comparator): Patients in the IR tacrolimus (Prograf) maintenance group will continue with their current dose of IR tacrolimus (Prograf) before enrollment unless the drug trough levels deviate from the therapeutic range.
  Interventions: Drug: Maintenance of immediate-release tacrolimus

INTERVENTIONS:
Drug: Conversion to extended-release tacrolimus — Conversion from immediate-release tacrolimus (Prograf) to extended-release tacrolimus (Envarsus XR) as a part of the maintenance immunosuppressive treatment
  Other Names: Envarsus XR
  Arms: Envarsus XR conversion
Drug: Maintenance of immediate-release tacrolimus — Continuing immediate-release tacrolimus (Prograf) as a part of the maintenance immunosuppressive treatment
  Other Names: Prograf
  Arms: Prograf maintenance

SUMMARY:
The objective of this randomized controlled study is to assess the neurocognitive outcomes between individuals using immediate-release (IR) tacrolimus (Prograf®) and those who were converted to extended-release tacrolimus (Envarsus XR) among older kidney transplant recipients (KTRs).

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed consent for participation in the study
* Patients who have regular outpatient follow-up at the Massachusetts General Hospital (MGH) transplant center
* ≥1 year since the latest kidney transplantation
* On IR tacrolimus as maintenance therapy
* At a stable therapeutic tacrolimus level (5-10 ng/ml) over the last ≥3 months
* Stable kidney function [<20% variability between the last two estimated glomerular filtration rate (eGFR)]
* Utilizing English or Spanish as the primary language

Exclusion Criteria:

* Dual organ transplantation
* Rejection within the last three months
* History of moderate to severe dementia (defined by Dementia Severity Rating Scale ≥19)
* History of Parkinson's disease
* Decompensated liver disease
* Active cancer
* Uncontrolled depression or anxiety
* Blindness
* Deafness
* Intellectual disabilities
* Pregnancy
* eGFR <15 mL/min/1.73 m2 at the time of enrollment
* Total bilirubin >3.0 mg/dL

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
The difference in changes of neurocognitive function in intermediate-term (Total cognition composite, standard score) | 12 month
  Neurocognitive functions will be assessed across multiple cognitive domains using the NIH toolbox-Cognitive battery (NIHTB-CB) version 3. The NIHTB-CB version 3 encompasses seven tests to assess attention, executive function, language, memory, and processing speed. The total cognition composite will be derived by averaging normalized scores. The results will be reported in Standard Scores [SS; mean of 100, standard deviation (SD) of 15] adjusting the age of the subject. The investigators will compare the changes in standard score from baseline between the two intervention groups.
The difference in changes of neurocognitive function in intermediate-term (Fluid composite, standard score) | 12 month
  The fluid composite score will be obtained using the NIH toolbox-Cognitive battery (NIHTB-CB) version 3, similarly as described above. The fluid cognition composite will be derived by averaging normalized scores. The results will be reported in Standard Scores [SS; mean of 100, standard deviation (SD) of 15] adjusting the age of the subject. The investigators will compare the changes in standard score from baseline between the two intervention groups.
The difference in changes of neurocognitive function in intermediate-term (Crystallized composite, standard score) | 12 month
  The crystallized composite score will be obtained using the NIH toolbox-Cognitive battery (NIHTB-CB) version 3, similarly as described above. The crystallized cognition composite will be derived by averaging normalized scores. The results will be reported in Standard Scores [SS; mean of 100, standard deviation (SD) of 15] adjusting the age of the subject. The investigators will compare the changes in standard score from baseline between the two intervention groups.
The difference in changes of neurocognitive function in intermediate-term (Total cognition composite, T score) | 12 month
  The total composite score will be obtained using the NIH toolbox-Cognitive battery (NIHTB-CB) version 3, similarly as described above. The total cognition composite will be derived by averaging normalized scores. The results will be reported in T scores (mean of 50 and SD of 10) with adjustments for age, gender, education, and race/ethnicity. The investigators will compare the changes in T score from baseline between the two intervention groups.
The difference in changes of neurocognitive function in intermediate-term (Fluid composite, T score) | 12 month
  The fluid composite score will be obtained using the NIH toolbox-Cognitive battery (NIHTB-CB) version 3, similarly as described above. The fluid cognition composite will be derived by averaging normalized scores. The results will be reported in T scores (mean of 50 and SD of 10) with adjustments for age, gender, education, and race/ethnicity. The investigators will compare the changes in T score from baseline between the two intervention groups.
The difference in changes of neurocognitive function in intermediate-term (Crystallized composite, T score) | 12 month
  The crystallized composite score will be obtained using the NIH toolbox-Cognitive battery (NIHTB-CB) version 3, similarly as described above. The crystallized cognition composite will be derived by averaging normalized scores. The results will be reported in T scores (mean of 50 and SD of 10) with adjustments for age, gender, education, and race/ethnicity. The investigators will compare the changes in T score from baseline between the two intervention groups.

SECONDARY OUTCOMES:
The difference in changes of neurocognitive function in short-term (Total cognition composite, standard score) | 3 month
  Same as described above
The difference in changes of neurocognitive function in short-term (Fluid composite, standard score) | 3 month
  Same as described above
The difference in changes of neurocognitive function in short-term (Crystallized composite, standard score) | 3 month
  Same as described above
The difference in changes of neurocognitive function in short-term (Total cognition composite, T score) | 3 month
  Same as described above
The difference in changes of neurocognitive function in short-term (Fluid composite, T score) | 3 month
  Same as described above
The difference in changes of neurocognitive function in short-term (Crystallized composite, T score) | 3 month
  Same as described above
The changes in quality of life, measured by SONG-LP questionnaire | 3 month and 12 month
  The Standardized Outcome in Nephrology-Life Participation (SONG-LP) questionnaire will evaluate each participant's engagement in significant life domains in correlation with the intervention. This questionnaire assesses life participation in the areas of leisure, family, work, and social activities through four simple questions. The score ranges from 4 to 20, with a higher score indicating greater engagement in life activities. The difference in changes of total score from baseline between the two intervention groups will be obtained.
The changes in tremor, measured by QUEST questionnaire | 3 month and 12 month
  Quality of Life in Essential Tremor (QUEST) questionnaire will be used to assess tremors subjectively. This questionnaire comprises 30 items contributing to the five dimensions: physical/activities of daily living, psychosocial, communication, hobbies/leisure, and work/finances. The investigators will also obtain self-rated tremor severity in various body parts. The score ranges from 0 to 120, with a higher score indicating a greater impact on their QOL from tremor. The investigators will compare the changes in total score and the score on each scale from baseline between the two intervention groups.
The changes in sleep quantity, measured by a wearable device | 3 month and 12 month
  The investigators will assess each participant's sleep quantity using wearable devices. The participants will be instructed to wear the device continuously for 14 days at pre-specified time points during the study period. Sleep quantity will be represented by the total amount of time spent asleep. The difference in changes in sleep quantity from baseline will be compared between the two intervention groups.
The changes in sleep quality, measured by a wearable device | 3 month and 12 month
  The investigators will objectively assess each participant's sleep quality using wearable devices. The participants will be instructed to wear the device continuously for 14 days at pre-specified time points during the study period. Sleep quality will be measured as a percentage of time spent in deep sleep and REM sleep to the total sleep time. A higher percentage indicates a better sleep quality. The changes in sleep quality from baseline will be compared between the two intervention groups.

OTHER OUTCOMES:
Subgroup analysis of primary and secondary outcomes based on age group | At 3 month and 12 month
  The investigators will analyze the differential impact of the intervention in participants aged 75 years and older, compared to those under 75 years old.
Subgroup analysis of primary and secondary outcomes based on gender | At 3 month and 12 month
  The investigators will perform a subgroup analysis for each outcome based on gender to determine whether the treatment effect varies between males and females.
Subgroup analysis of primary and secondary outcomes based on education level | At 3 month and 12 month
  The investigators will analyze the differential impact of the intervention in participants with Bachelor's degree holders, compared to those without Bachelor's degree holders.
Subgroup analysis of primary and secondary outcomes based on the baseline cognitive function | At 3 month and 12 month
  The investigators will perform a subgroup analysis for each outcome based on baseline cognitive function to determine whether the treatment effect varies according to baseline cognitive function. Participants with a baseline NIHTB-CB total composite T score ≤ 43 (corresponding to the lower 25th percentile adjusted for age, gender, education, and race/ethnicity) will be separately analyzed to those with a score > 43.

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo V. Riella, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- MGH Kidney Transplant Clinic, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
As part of our commitment to transparency and promoting further scientific research, the investigators plan to share individual participant data (IPD) from this clinical trial. The data will be made available to qualified researchers upon request, subject to appropriate data use agreements and ethical considerations. Specifically, the following data will be shared:
  Demographic Information: Age, sex, race. Outcomes Data: Information related to primary and secondary endpoints Adverse Events: Data on reported adverse events and serious adverse events.
  All data will be available in a de-identified format to protect participant confidentiality via ClinicalTrials.gov.
Supporting Information: Study Protocol
Time Frame: The individual participant data (IPD) and supporting information will be made available to qualified researchers 6 months after the publication of the primary study results. Data will be accessible for a minimum of 5 years from the date of publication or study completion, whichever occurs later, to ensure ample time for further research and analysis.
Access Criteria: Access to individual participant data (IPD) will be granted to qualified researchers conducting non-commercial, scientifically valid research. Researchers must:
  1. Submit a formal data access request, including a research proposal and ethical review approval.
  2. Sign a data use agreement outlining the terms of data use, including confidentiality and non-re-identification.
  3. Provide documentation of ethical approval from an Institutional Review Board or equivalent.